CLINICAL TRIAL: NCT04555850
Title: A Randomized, Double-blind, Placebo-Controlled, Multiple Doses,Dose-escalation，Phase 1b Study of the Safety, Tolerability，Pharmacokinetics and the Potential Immunological Reaction of Recombinant Human Thymosin Beta4 in Chinese Healthy Volunteers
Brief Title: A Phase 1b Study of Thymosin Beta 4 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL005-Ⅰ-2015-2
Record Dates: First submitted 2020-05-08; First posted 2020-09-21 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Recombinant human thymosin β4

STUDY DESIGN:
Intervention Model Description: Dose Escalation for 3 Cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Recombinant Human Thymosin β4 0.5ug/kg (Experimental): 10 subjects in this group will receive NL005 for 0.5ug/kg respective.Continuous administration for 10 days.
  Interventions: Drug: Recombinant Human Thymosin β4
- Recombinant Human Thymosin β4 2.0ug/kg (Experimental): 10 subjects in this group will receive NL005 for 2.0ug/kg respective.Continuous administration for 10 days.
  Interventions: Drug: Recombinant Human Thymosin β4
- Recombinant Human Thymosin β4 5.0ug/kg (Experimental): 10 subjects in this group will receive NL005 for 5.0ug/kg respective.Continuous administration for 10 days.
  Interventions: Drug: Recombinant Human Thymosin β4
- Placebo (Other): Two subjects in each dose group (0.5/2/5ug/kg) were given placebo for 10 days.A total of six participants were given a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Recombinant Human Thymosin β4 — Healthy subjects , were given a dose of rh-Tβ4 for ten consecutive days.
  Other Names: rh-β4
  Arms: Recombinant Human Thymosin β4 0.5ug/kg; Recombinant Human Thymosin β4 2.0ug/kg; Recombinant Human Thymosin β4 5.0ug/kg
Other: Placebo — 3 cohorts, with 6 healthy subjects , were given a dose of Placebo for ten consecutive days. Cohorts received ascending doses of either 0.5,2.0 or 5.0 ug/kg .
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerance, pharmacokinetics and the potential immunological reaction of single intravenous recombinant human thymosin β4（NL005）or placebo 0.5, 2.0,5.0μg/kg in Chinese healthy volunteers.30 volunteers will be randomly assigned to one of three groups to receive either NL005 or placebo for 10 consecutive days.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability pharmacokinetics and potential immune responses of multiple NL005 intravenous administration.

Three groups of 30 subjects will receive an NL005 or placebo dose of 0.5μg/kg 2.0 μg/kg and 5.0 μg/kg for 10 consecutive days at a ratio of 4:1.

While observing the safety of the subjects in each dose group, about 5mL of venous blood was collected for the ADA study in healthy subjects 14 days and 28 days after the first administration of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy volunteers（male or female）.
2. Between 18 and 50 years of age.
3. Female subjects should weigh no less than 45 kg and male subjects should weigh no less than 50 kg.BMI between 19 and 28 kg/m2.
4. Good health condition, no history of unintentional, liver, kidney, digestive tract, immune system, nervous system, mental and metabolic abnormality, no family history of tumor.
5. Ability to communicate normally with medical staff, understand research requirements and comply with hospital regulations.
6. Voluntarily sign informed consent.

Exclusion Criteria:

1. Physical examination vital signs electrocardiogram and laboratory examination are not done or any result is judged to be clinically significant abnormal (judged by clinician).
2. ADA tests positive.
3. Smoking more than 5 cigarettes a day for the previous 3 months, or no guarantee to stop smoking during the trial.
4. Previous history of substance abuse or drug screening test positive.
5. Alcohol intake averaged more than 2 units per day (1 unit = 360mL beer,150mL wine or 45mL 40% alcohol liquor) or alcohol test positive in the first 3 months of inclusion.
6. Participated in another trial or used this drug within 3 months before inclusion.
7. Any other drug was used within two weeks before the trial.
8. There is a significant clinical history of allergy, especially for drugs, protein preparations and biological products, especially for rh-tβ4 or any of its ingredients.
9. Blood donation or blood loss was equal to or greater than 400 mL within three months prior to the trial.
10. Female subjects who are pregnant or breast-feeding, or who are likely to become pregnant without using an acceptable method of contraception, or who are positive for a pregnancy test, and male subjects who are not using effective contraception or whose partner has a family planning plan within six months of the end of the trial.
11. Unable to tolerate venous blood collection.
12. There is no guarantee that smoking and taking grapefruit juice or any alcoholic and xanthine food and beverage (including chocolate, tea, coffee, cola, etc.) from 48 hours before administration to the last blood sample collection.
13. The investigator judges that the subject is unable to complete the study or otherwise considers that the subject's participation in the study may cause other injury.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) . | Day-7、-1、1、2、3、4、5、6、7、8、9、10、14、28.
  Determine maximum tolerated dose (MTD) or dose-limiting toxicity (DLT) by comprehensive evaluation of drug safety by adverse event observation, vital signs, physical examination, laboratory examination, electrocardiogram, etc. In this study, DLT was defined as liver, kidney, heart and mental nervous system toxicity of level 2 or above or blood system toxicity of level 3 or above and other systemic adverse events occurred within 14 days after drug administration, and the adverse events were judged to be related to the experimental drug use.If more than 3 (including 3) DLT cases are present in any dose group, the test should be terminated. The previous dose of this dose is considered the maximum tolerated dose (MTD).
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. | Day-7、-1、1、2、3、4、5、6、7、8、9、10、14、28.
  Determine maximum tolerated dose (MTD) or dose-limiting toxicity (DLT) by comprehensive evaluation of drug safety by adverse event observation, vital signs, physical examination, laboratory examination, electrocardiogram, etc. All adverse events were determined according to NCI CTCAE4.03.CTCAE4.03 was classified into grades 1 to 5, in which grade 1 was mild adverse event and grade 5 was death due to adverse event.According to NCI CTCAE4.03.
The Cmax of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The Tmax of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The MRT of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The AUClast of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The AUC0-inf of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The t1/2 of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The VZ of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The CL of multiple administration of rh-Tβ4. | Day 1、2、3、4、5、6、7、8、9、10.
  Approximately 5mL of venous blood was collected at allotted time for the pharmacokinetic study of rh-Tβ4 in healthy subjects for the prescribed time.The pharmacokinetic parameters included Cmax , tmax ,MRT ,AUClast ,AUC0-inf,t1/2 ,VZ , CL.
The potential immunological reaction (antibody formation) of multiple administration of rh-Tβ4. | Day 1、14、28.
  Approximately 5mL venous blood was collected from subjects before, 14 days after, and 28 days after administration for ADA study of rh-Tβ4 in healthy subjects.After the 28th-day follow-up period, subjects who confirm that ADA results are positive should be reexamined every 30 days (±3 days) until the results turn negative or the titer level is stable for two consecutive times.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Beijing, China

REFERENCES:
- See also: Related Info — http://www.northland-bio.com/